CLINICAL TRIAL: NCT00280501
Title: Dopaminergic Modulation of Choroidal Blood Flow Changes During Dark/Light Transitions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjaeger-Mayrl, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-160905
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Regional Blood Flow; Ocular Physiology
Keywords: Sulpiride; Quetiapine; Light/dark transition; Choroidal blood flow
MeSH Terms: interventions — Quetiapine Fumarate; Pharmaceutical Preparations; Sulpiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Quetiapine
  Interventions: Drug: Quetiapine (drug); Drug: Sulpiride (drug); Drug: Placebo
- 2 (Active Comparator): Sulpiride
  Interventions: Drug: Quetiapine (drug); Drug: Sulpiride (drug); Drug: Placebo
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Quetiapine (drug); Drug: Sulpiride (drug); Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine (drug) — Quetiapine (Seroquel 100mg-film-coated tablet, AstraZeneca Vienna, Austria) Dose: 100 mg tablet oral single dose
Drug: Sulpiride (drug) — Sulpiride (Dogmatil 200mg-tablet, Synthélabo Groupe, Le Plessis Robinson, France) Dose: one half of 200 mg tablet oral single dose
Drug: Placebo — Placebo

SUMMARY:
There is evidence from a variety of animal studies that choroidal blood flow is under neural control. By contrast, only little information is available from human studies. Recent results indicate that a light/dark transition is associated with a reduction in choroidal blood flow due to an unknown mechanism. We have shown that during unilateral dark/light transitions both eyes react with choroidal vasoconstriction strongly indicating a neural mechanism responsible for the blood flow changes.

Dopamine has been discussed as a chemical messenger for light adaptation. However, dopaminergic effects in the eye are not restricted to synaptic sites of release, but dopamine also diffuses to the outer retinal layers and pigment epithelium. Accordingly, dopaminergic effects also include a modulatory role on retinal vessel diameter and animal studies provide evidence for vasodilatory effects in the choroid. There is evidence that during darkness retinal and choroidal dopamine levels decrease. Accordingly, dopamine could provide a modulatory input to the light/dark transition induced changes of choroidal circulation. The aim of the present study is to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
choroidal blood flow | in total 3x 3 hours
fundus pulsation amplitude | in total 3 x 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria